CLINICAL TRIAL: NCT06885996
Title: Psilocybin-assisted Therapy for Post-Traumatic Stress Disorder in Survivors of Intimate Partner Violence
Acronym: PsiPTSD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Vancouver Island University (Unknown); University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB25-0065
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-02

CONDITIONS: Post Traumatic Stress Disorder PTSD; Intimate Partner Violence (IPV)
Keywords: Psychotherapy; Psilocybin; Acceptance and Commitment Therapy
MeSH Terms: conditions — Combat Disorders | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The group assignments to active (high dose) and control (low dose) psilocybin-assisted therapy will be based on a blocked randomization list (10 participants per block) using sealed envelopes created by an employee of the University of Calgary, who will not be involved in the conduct, or the analysis of the study.
  The pharmacies administering the psilocybin will be responsible for maintaining the master randomization code list and only the technician preparing the samples will have access to the envelopes and code list.
  When a new study ID is generated, the technician is to verify the randomization and prepare the participant's study intervention accordingly. Unblinding will only occur once the entire study is completed, and the database has been locked.
  The trials active intervention and comparator will be provided by the manufactures and will be identical in shape, colour, and weight.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Dose (Experimental): High Dose (25mg) PEX010 (Oral Psilocybin), 25mg; single dose (38 participants) administered 24hrs prior to first ACT session
- Low Dose (Active Comparator): Low Dose (1mg) PEX010 (Oral Psilocybin), 1mg; single dose (20 participants) administered 24hrs prior to first ACT session
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — See treatment arm description.
  Arms: Low Dose

SUMMARY:
The goal of this randomized controlled trial is to evaluate the efficacy of psilocybin administered with Acceptance and Commitment Therapy (ACT) as an intervention to reduce post-traumatic stress disorder (PTSD) symptom burden in adult (aged 18-65) survivors of intimate partner violence (IPV).

This trail will test the following 2 aims:

AIM 1 : To compare the efficacy of a therapeutic psilocybin dose at improving outcomes on the PCL-5 and CAPS-5 as compared to an active control psilocybin dose in IPV survivors with chronic PTSD.

AIM 2: To evaluate the efficacy of psilocybin on quality of life, cognitive function, motor ability, depression, anxiety, and cognitive flexibility.

Participants will be asked to:

* Complete a 2 part screening process
* Attend a baseline assessment
* Complete a psychoeducation preparation session(s)
* Attend psilocybin administration session (receive high dose [25mg] or low dose psilocybin [1mg])
* Complete 5-6 weekly sessions of ACT
* Repeat outcome measures at 1-week, 4 weeks, 3 months (online questionnaires only), and 6 months post-psilocybin administration.

DETAILED DESCRIPTION:
The overall objective of this study is to evaluate the efficacy of psilocybin administered with Acceptance and Commitment Therapy (ACT) as an intervention to reduce post-traumatic stress disorder (PTSD) symptom burden in survivors of intimate partner violence (IPV).

This trail will test the following 2 aims:

AIM 1 : To compare the efficacy of a therapeutic psilocybin dose (25mg) at improving outcomes on the PCL-5 and CAPS-5 as compared to an active control psilocybin dose (1mg) (allocation ratio 1:1) in IPV survivors with chronic PTSD. Mean baseline scores will be compared to scores at each follow-up timepoint (1-week, 4 weeks, 3 months (PCL-5 only), and 6 months post-psilocybin administration).

AIM 2: to evaluate the efficacy of psilocybin on quality of life, cognitive function, motor ability, depression, anxiety, and cognitive flexibility. Mean baseline scores will be compared to scores at each follow-up timepoint (1-week, 4 weeks, 3 months (online only), and 6 months post-psilocybin administration).

The secondary efficacy outcomes will include measures of mood, anxiety, post-traumatic stress, cognitive flexibility, emotional regulation, and quality of life.

Exploratory Aim: Exploratory objectives of this study include evaluating blood biomarkers reflective of inflammation, growth factors, brain injury, and oxidative stress relevant to PTSD and psilocybin's mechanisms of action.

A total of 76 male and female patients between the ages of 18-65 with the last incident of IPV greater than 6 months prior with a score of 1 on the Composite Abuse Scale with repetition of abusive events, meeting DSM-5 criteria for PTSD and a minimum PCL-5 score of 33.

All patients will undergo a thorough, 2-part screening procedure. Eligible participants will be randomly allocated 1:1 to either the high dose (38 participants) or low dose (38 participants) psilocybin groups. All participants will be asked to attend a baseline session consisting of clinical and behavioural outcome measures followed by a pre-dosing psychoeducation session. Following the single dosing session, participants will complete 5-6 weekly ACT sessions. Outcome measure assessments will be repeated at 1-week, 4 weeks, 3 months (online only), and 6 months post-dosing.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of all sexes, gender identities, and ethnicities
* Ages 19 to 65 years at the time of screening
* At least 6 months since last IPV incident
* A score of 1 on the Composite Abuse Scale with repetition of abusive events
* Minimum PCL-5 score of ≥ 33
* Limited lifetime use of serotonergic hallucinogens
* Ability to read/write English

Exclusion Criteria:

* Severe or moderate substance use disorder other than nicotine in past 6 months
* Lifetime diagnosis of schizophrenia or bipolar disorders (or first or second-degree relative)
* Active suicidal ideation or serious attempt within the past 1 year.
* Current pregnancy or nursing, trying to become pregnant
* Any notable abnormality on ECG or routine medical blood laboratory test
* Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia
* Epilepsy with a history of seizures
* Current or recent (within 12 weeks) participation in a clinical trial
* Cognitive impairment (SLUMS score <20)
* Suffered a moderate/severe TBI at least once in lifetime
* Suffered a mild TBI within the last 6 months
* Any other circumstances that, in the opinion of the investigators, compromises participant safety
* Not compelled to enter treatment to avoid legal consequences

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | Change from baseline to 1-week, 4 weeks, and 6 months post-dosing
  A clinician-administered, 30-item structured interview to diagnose and assess severity of PTSD symptoms in patients. It is widely used and validated, and is considered the gold standard PTSD diagnostic tool.
PTSD Checklist for DSM-5 (PCL-5) | Change from baseline to 1-week, 4 weeks, and 3 months, and 6 months post-dosing
  A 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD.

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale, Self-Reported (MADRS-S) | Change from baseline to 1-week, 4 weeks, 3 months, and 6 months post-dosing
  A self-reported, 9-item assessment of depressive symptoms using a recall period of the past 7 days. This tool elicits a total score ranging from 0-54, with higher scores indicating greater depression.
Generalized Anxiety Disorder-7 (GAD-7) | Change from baseline to 1-week, 4 weeks, and 3 months, and 6 months post-dosing
  A 7-item self-reported questionnaire for measuring the severity of generalized anxiety disorder. Individuals rate how often they have been bothered by seven listed problems and score their responses from 0 ("not at all") to 3 ("nearly every day"). Total scores for anxiety severity are: 0-4: minimal anxiety; 5-9: mild; 10-14: moderate; 15-21: severe anxiety
Rivermead Post-Concussion Symptoms Questionnaire (RPQ) | Change from baseline to 1-week, 4 weeks, and 3 months, and 6 months post-dosing
  A self-reported, 16-item questionnaire used to assess severity of 16 commonly experienced PPCS symptoms using a scale of 0 ("not experienced") to 4 ("severe problem"), with higher scores indicating greater PPCS symptom burden.
The Acceptance and Action Questionnaire II (AAQ-II) | Change from baseline to 1-week, 4 weeks, and 6 months post-dosing
  A 7-item questionnaire measuring psychological flexibility. Scores range from 0 to 49 with higher scores indicating greater psychological flexibility.
Cognitive Fusion Questionnaire (CFQ-7) | Change from baseline to 1-week, 4 weeks, and 6 months post-dosing
  A 7-point Likert scale measuring cognitive fusion. Scores range from 0 to 49 with higher scores indicating greater fusion with one's thoughts.
The Sheehan Disability Scale (SDS) | Change from baseline to 1-week, 4 weeks, and 6 months post-dosing
  A three-part, self-reported rating of functional impairment in the three major life domains: work, home and social life, and family responsibilities. Total scores range from 0 to 30 and aim to identify how symptoms have disrupted these life domains.
9. EuroQol-5D (EQ-5D-5L) | Change from baseline to 1-week, 4 weeks, and 6 months post-dosing
  A self-report measure of 5 key life dimensions, designed to measure health-related quality of life.
Cognitive Flexibility Scale (CFS) | Change from baseline to 1-week, 4 weeks, and 6 months post-dosing
  A 12-item Likert-scale designed to assess the ability to identify options and alternatives to a situation, flexibility in behaviour, and confidence in the flexible behaviour.
The Trail-Making Test 'B' (TMT-B) | Change from baseline to 1-week, 4 weeks, and 6 months post-dosing
  The Trail-Making Test 'B' (TMT-B) is a test of general cognitive function, designed to assess working memory, visual processing, visuospatial skills, selective and divided attention, processing speed, and psychomotor coordination. The measure for this 3 to 4-min task is the time required for accurate completion
The Digit Span Task (DS) | Change from baseline to 1-week, 4 weeks, and 6 months post-dosing
  The Digit Span Task (DS)is a measure of verbal short term and working memory designed to measure simple attention. This 1 to 3-min task required participants to repeat a series of digits increasing in length and is measured through direction of the task, longest sequence successfully complete, and total number of attempts.
The Rey Auditory Verbal Learning Test (RAVLT) | Change from baseline to 1-week, 4 weeks, and 6 months post-dosing
  The Rey Auditory Verbal Learning Test (RAVLT) is a neuropsychological assessment that evaluates memory dysfunction by examining short-term auditory-verbal memory, learning rate and strategies, interference effects, confabulation, information retention, and learning-retrieval differences.
Symbol Digit Modalities Test (SDMT) | Change from baseline to 1-week, 4 weeks, and 6 months post-dosing
  The Symbol Digit Modalities Test (SDMT) is a neuropsychological test used to assess information processing speed and cognitive function, particularly in individuals with neurological disorders like multiple sclerosis. It involves matching symbols to numbers within a 90-second time limit.

OTHER OUTCOMES:
Blood biomarkers | Change from baseline to 1-week, 4 weeks, and 6 months post-dosing
  To explore blood biomarkers related to PTSD, brain injury, inflammation, oxidative stress, and growth factors following psilocybin-assisted therapy

CONTACTS AND LOCATIONS:
Overall Officials: Sandy Shultz, PhD, Principal Investigator — Director, Centre for Trauma and Mental Health Research, Vancouver Island University; Leah Mayo, PhD, Principal Investigator — Parker Psychedelics Research Chair and Assistant Professor, Department of Psychiatry, University of Calgary, Cumming School of Medicine; Pamela Kryskow, MD, CCFP, Principal Investigator — Medical Lead, Psychedelic-assisted Therapy Graduate Program, Vancouver Island University, Medical Director, Roots to Thrive Society; Zachary Walsh, PhD, Principal Investigator — Professor, Department of Psychology, University of British Columbia; Paul van Donkelaar, PhD, Principal Investigator — Professor, Faculty of Health and Social Development, School of Health and Exercise Sciences; Shannon Dammes, RN, MPH, Principal Investigator — Professor, Health Sciences, Vancouver Island University, and Visioning and Development Lead, Roots to Thrive Society; Jodie Gawryluk, PhD, Principal Investigator — Associate Professor, Department of Psychology, University of Victoria
Locations (3):
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - The University of British Columbia - Okanagan Campus, Kelowna, British Columbia
  - Vancouver Island University, Nanaimo, British Columbia

IPD SHARING:
Plan to Share IPD: No